CLINICAL TRIAL: NCT04878653
Title: Alcohol-Containing Products' Effect on Breathalyzer Results in Healthy Adults Without Acute Intoxication
Status: Completed | Type: Observational
Sponsor: CHRISTUS Health (Other)
Responsible Party: Principal Investigator, Jordyn Ewbank, DO, Principal Investigator, CHRISTUS Health
Other Study IDs: 2019-106
Record Dates: First submitted 2020-11-25; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Alcohol Drinking; Intoxication Alcohol
MeSH Terms: conditions — Alcohol Drinking; Alcoholic Intoxication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: BACtrack S80 Breathalyzer — The breathalyzer, BACtrack S80 Breathalyzer, will be calibrated per manufacturer's recommendations before each reading will be taken. Participants will administer the breathalyzer test on themselves. They will be instructed on how to hold and blow into the breathalyzer machine.

SUMMARY:
This study is a prospective, controlled study in healthy volunteers all of whom are residents, medical students, faculty physicians, or emergency department nursing and ancillary staff.

DETAILED DESCRIPTION:
The breathalyzer, BACtrack S80 Breathalyzer, will be calibrated per manufacturer's recommendations before each reading will be taken. Participants will administer the breathalyzer test on themselves. They will be instructed on how to hold and blow into the breathalyzer machine. Participants will then be instructed to wash his or her hands and an initial breathalyzer reading will be taken and will serve as the control prior to the application of each product. Participants with a result >0 will be excluded from the study. Participants will apply the alcohol-containing product to his or her hands and a second breathalyzer reading will be obtained immediately after application. If the second breathalyzer result is >0, a third breathalyzer reading will be obtained after the product has dried appropriately on the participant's hands (approximately 1 minute after initial application). A minimum of two breathalyzer readings will be obtained from each participant per product application. If the second breathalyzer reading is >0, a third breathalyzer will be obtained from that participant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals between the ages of 18 and 75
* Able to verbally consent
* Residents, medical students, faculty physicians, emergency department nursing and ancillary staff

Exclusion Criteria:

* Inability to consent
* Individuals with an initial breathalyzer result greater than 0.000
* Individuals who have consumed alcohol or used other alcohol-containing products within the last 12 hours

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A maximum of 50 healthy individuals between the ages of 18 and 75 who are willing to participate and able to verbally consent for this study. Volunteers will include residents, medical students, faculty physicians, or emergency department nursing and ancillary staff. Demographics collected for each participant will include age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-10-22 (Actual); Study Completion 2020-10-22 (Actual)

PRIMARY OUTCOMES:
Patient breath alcohol concentration (BrAC) | Through study completion, an estimate of 6 months
  1. The BACtrack S80 Breathalyzer was used in this study to measure each individual's breath alcohol concentration (BrAC) to estimate one's blood alcohol concentration (BAC). It is measured as a percentage, i.e. a measurement of 0.040 represents 0.04%. The generally accepted legal standard for alcohol intoxication in the United States is 0.08%. The Outcome Measures include mean readings for each group looking at readings greater than 0%, greater than 0.04%, and greater than 0.08%.

CONTACTS AND LOCATIONS:
Overall Officials: Jordyn Ewbank, DO, Principal Investigator — CHRISTUS Health
Locations (1):
- CHRISTUS Spohn Hospital, Corpus Christi, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Investigator is interested in pursuing future collaborations and grant opportunities.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Background] Klein LR, Cole JB, Driver BE, Battista C, Jelinek R, Martel ML. Unsuspected Critical Illness Among Emergency Department Patients Presenting for Acute Alcohol Intoxication. Ann Emerg Med. 2018 Mar;71(3):279-288. doi: 10.1016/j.annemergmed.2017.07.021. Epub 2017 Aug 24. PMID 28844504
- [Background] Sebbane M, Claret PG, Jreige R, Dumont R, Lefebvre S, Rubenovitch J, Mercier G, Eledjam JJ, de la Coussaye JE. Breath analyzer screening of emergency department patients suspected of alcohol intoxication. J Emerg Med. 2012 Oct;43(4):747-53. doi: 10.1016/j.jemermed.2011.06.147. Epub 2012 Mar 8. PMID 22406024
- [Background] Kumar A, Holloway T, Cohn SM, Goodwiler G, Admire JR. The Clinical Evaluation of Alcohol Intoxication Is Inaccurate in Trauma Patients. Cureus. 2018 Feb 14;10(2):e2190. doi: 10.7759/cureus.2190. PMID 29662729
- [Background] Phillips DP, Brewer KM. The relationship between serious injury and blood alcohol concentration (BAC) in fatal motor vehicle accidents: BAC = 0.01% is associated with significantly more dangerous accidents than BAC = 0.00%. Addiction. 2011 Sep;106(9):1614-22. doi: 10.1111/j.1360-0443.2011.03472.x. Epub 2011 Jun 20. PMID 21689195
- [Background] Ali SS, Wilson MP, Castillo EM, Witucki P, Simmons TT, Vilke GM. Common hand sanitizer may distort readings of breathalyzer tests in the absence of acute intoxication. Acad Emerg Med. 2013 Feb;20(2):212-5. doi: 10.1111/acem.12073. PMID 23406081
- [Background] Foglio-Bonda PL, Poggia F, Foglio-Bonda A, Mantovani C, Pattarino F, Giglietta A. Determination of breath alcohol value after using mouthwashes containing ethanol in healthy young adults. Eur Rev Med Pharmacol Sci. 2015;19(14):2562-6. PMID 26221882
- [Background] Modell JG, Taylor JP, Lee JY. Breath alcohol values following mouthwash use. JAMA. 1993 Dec 22-29;270(24):2955-6. PMID 8254857
- [Background] Lindsay HA, Hannam JA, Bradfield CN, Mitchell SJ. Breath alcohol of anesthesiologists using alcohol hand gel and the "five moments for hand hygiene" in routine practice. Can J Anaesth. 2016 Aug;63(8):938-44. doi: 10.1007/s12630-016-0666-2. Epub 2016 May 3. PMID 27142004
- [Background] Strawsine E, Lutmer B. The Effect of Alcohol-Based Hand Sanitizer Vapors on Evidential Breath Alcohol Test Results. J Forensic Sci. 2018 Jul;63(4):1284-1290. doi: 10.1111/1556-4029.13691. Epub 2017 Nov 16. PMID 29143333
- [Background] Freudenrich C. How breathalyzers work. https://electronics.howstuffworks.com/gadgets/automotive/breathalyzer.htm . Updated October 20, 2000. Accessed February 2, 2019.
- [Background] Duke University. The alcohol pharmacology education partnership. https://sites.duke.edu/apep/module-4-alcohol-and-the-breathalyzer-test/. Accessed February 2, 2019.
- [Background] Labianca, DA. The flawed nature of the calibration factor in breath-alcohol analysis. J Chemical Edu. 2002;79(10):1237-1240.
- [Background] Caravati EM, Anderson KT. Breath alcohol analyzer mistakes methanol poisoning for alcohol intoxication. Ann Emerg Med. 2010 Feb;55(2):198-200. doi: 10.1016/j.annemergmed.2009.07.021. Epub 2009 Oct 14. PMID 19833410
- [Background] Arndt T, Schrofel S, Gussregen B, Stemmerich K. Inhalation but not transdermal resorption of hand sanitizer ethanol causes positive ethyl glucuronide findings in urine. Forensic Sci Int. 2014 Apr;237:126-30. doi: 10.1016/j.forsciint.2014.02.007. Epub 2014 Feb 18. PMID 24631832
- [Background] Arndt T, Gruner J, Schrofel S, Stemmerich K. False-positive ethyl glucuronide immunoassay screening caused by a propyl alcohol-based hand sanitizer. Forensic Sci Int. 2012 Nov 30;223(1-3):359-63. doi: 10.1016/j.forsciint.2012.10.024. Epub 2012 Nov 5. PMID 23137849